CLINICAL TRIAL: NCT07309757
Title: Maternal Outcomes With Methamphetamine Use and Cardiac Assessment for Rural Dissemination (MOM CARD)
Status: Not yet recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Evan Shalen, Assistant Professor, Oregon Health and Science University
Other Study IDs: STUDY00028946
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Methamphetamine Abuse
Keywords: Methamphetamine use; Pregnancy; Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to develop a pilot screening protocol, comparing cardiac point-of-care ultrasound (POCUS), electrocardiogram (EKG), serum biomarkers (N-terminal pro b-type natriuretic peptide (NT-proBNP), high sensitivity troponin (hsTn)) with formal transthoracic echocardiogram (TTE) in pregnant women with methamphetamine use.

DETAILED DESCRIPTION:
This is a pilot study that examines previously undiagnosed cardiac pathology utilizing transthoracic echocardiogram (TTE) in pregnant women with chronic methamphetamine use and assesses possible screening modalities (cardiac point-of-care ultrasound (POCUS), serum biomarkers, electrocardiogram (EKG)) in identifying underlying disease in this population. As this is a prospective observational study, we will assess pregnancy-related complications and care connections in the pilot tertiary academic setting.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older > 20 weeks gestation admitted to the hospital
* Active patient-defined regular methamphetamine use for at least 1 year and any use within the last month
* Able to understand and provide informed consent
* Able to understand English

Exclusion Criteria:

These criteria will exclude women whose medications, personal traits, obstetric conditions, or diseases could confound cardiovascular risk.

* Prescribed stimulants
* Echocardiogram or EKG previously performed during current pregnancy
* Previous diagnosis of congestive heart dysfunction
* Previous diagnosis of pulmonary hypertension
* Previous myocardial infarction
* Previous diagnosis of endocarditis
* Prior cardiac intervention (repair of cardiac congenital lesion, valve replacement or repairs, percutaneous/operative treatment of arrhythmias)
* High-risk aortopathy (Marfan syndrome, bicuspid aortopathy, prior aortic dissection)

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Pregnant women > or equal to 20 weeks gestation presenting to OHSU for hospital, day patient, or observation admission will be identified via the electronic medical record.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of point of care cardiac ultrasound for the detection of left ventricular systolic dysfunction as compared to comprehensive transthoracic echocardiogram. | Day 1
  This outcome seeks to identify the sensitivity of point of care cardiac ultrasound for the identification of left ventricular systolic dysfunction in pregnant people who use methamphetamine when performed by an obstetrics provider, as compared to formal transthoracic echocardiogram.

SECONDARY OUTCOMES:
Sensitivity of cardiac biomarkers and ECG for the identification of left ventricular systolic dysfunction as compared to comprehensive transthoracic echocardiogram. methamphetamine | Day 1
  This outcome seeks to identify the sensitivity of N-terminal pro-B-type natriuretic peptide (NT-proBNP), high sensitivity troponin and electrocardiogram for the identification of left ventricular systolic dysfunction in pregnant people who use methamphetamine, as compared to formal transthoracic echocardiogram.
Prevalence of underlying structural heart disease in pregnant people who use methamphetamine | Day 1
  This outcome seeks to identify the prevalence of structural heart disease in pregnant people who use methamphetamine.
Pregnancy and delivery outcomes in people who use methamphetamine | 3 months postpartum
  This outcome seeks to identify the prevalence of pregnancy delivery complications in people who use methamphetamine.
Changes to pregnancy-related treatment plan based on cardiovascular screening in people who use methamphetamine. | 3 months postpartum
  This outcome seeks to identify linkage to cardiovascular and addiction specialty care among patients diagnosed with cardiovascular disease.

IPD SHARING:
Plan to Share IPD: No